CLINICAL TRIAL: NCT01354470
Title: A Randomized, Placebo-Controlled Trial of Modafinil for Methamphetamine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Responsible Party: Principal Investigator, Gantt Galloway, PharmD, Scientist, California Pacific Medical Center Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPMC-APRL-8B
Record Dates: First submitted 2011-05-12; First posted 2011-05-17 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Methamphetamine Dependence
Keywords: Meth; Methamphetamine Addiction; Methamphetamine Treatment; Modafinil
MeSH Terms: interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Modafinil (Experimental)
  Interventions: Drug: Modafinil
- placebo (cornstarch) (Placebo Comparator)

INTERVENTIONS:
Drug: Modafinil — 600 mg Modafinil capsule
  Arms: Modafinil

SUMMARY:
The proposed study will establish the safety and efficacy of modafinil in the treatment of methamphetamine dependence, as well as assess the affects of modafinil on cognitive function in methamphetamine users and on methamphetamine withdrawal symptoms. In this outpatient trial, methamphetamine- dependent, treatment-seeking subjects will receive modafinil or placebo daily for four weeks, along with weekly Motivational Enhancement Therapy sessions. This study will be conducted at the Addiction & Pharmacology Laboratory in San Francisco, CA, and at the New Leaf Treatment Center in Lafayette, CA, and is expected to last one year.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years
* Patient is agreeable to conditions of study and signs consent form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Urine Samples Negative for Methamphetamine | Twice weekly for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gantt Galloway, PharmD, Principal Investigator — California Pacific Medical Center
Locations (2):
- United States (2):
  - New Leaf Treatment Center, Lafayette, California
  - CPMC Research Institute, St.Luke's Hospital, San Francisco, California